CLINICAL TRIAL: NCT05132361
Title: A Prospective Randomized Multicenter Single Blinded Study to Assess the Safety and Efficacy of the SELUTION SLR™ 018 Drug Eluting Balloon in the Treatment of Subjects With Femoropopliteal Artery Lesions
Brief Title: SELUTION4SFA Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.A. Med Alliance S.A. (Industry)
Collaborators: NAMSA (Other); Cordis US Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S2020-02
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-06

CONDITIONS: Peripheral Arterial Disease; Superficial Femoral Artery Stenosis
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Angioplasty, Balloon

STUDY DESIGN:
Who Masked: Participant
Masking Description: The physician performing the index procedure as well as study site personnel present at the index procedure will not be blinded, however, every effort will be made to maintain blinding for the following:
  * Subjects and their families
  * Site personnel only involved in conducting study assessments during follow-up.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- SELUTION SLR™ 018 DEB (Experimental): Treatment with Selution SLR drug eluting balloon to apply long term (>90 days) local treatment with sirolimus
  Interventions: Device: SELUTION SLR™ 018 DEB
- Plain (Uncoated) Balloon Angioplasty (PTA) (Active Comparator): Opening artery only by dilatation with an temporary inserted and inflated balloon.
  Interventions: Device: Plain (Uncoated) Balloon Angioplasty (PTA)

INTERVENTIONS:
Device: SELUTION SLR™ 018 DEB — a non-surgical procedure that uses a catheter to inflate a drug-eluting balloon to open up above the-knee arteries that have been narrowed due to peripheral arterial disease.
  Arms: SELUTION SLR™ 018 DEB
Device: Plain (Uncoated) Balloon Angioplasty (PTA) — a non-surgical procedure that uses a catheter to inflate a commercially available, non-drug-eluting balloon to open up above the-knee arteries that have been narrowed due to peripheral arterial disease.
  Arms: Plain (Uncoated) Balloon Angioplasty (PTA)

SUMMARY:
This study aims to demonstrate the safety and efficacy of the SELUTION SLR™ 018 DEB compared to plain (uncoated) balloon angioplasty in the treatment of peripheral arterial disease (PAD) in the superficial femoral artery (SFA) and proximal popliteal artery (PPA).

DETAILED DESCRIPTION:
Prospective, multi-center, single blinded, 2:1 randomized, controlled, superiority clinical trial.

This study will enroll up to 300 randomized subjects, and up to 20 subjects in a parallel pharmacokinetic (pK) sub study, at up to 60 clinical sites in the United Stated (US), Europe (EU) and Asia. A minimum of 50% of randomized subjects will be enrolled in the US. No more than 45 subjects (15% of the total randomized cohort) can be enrolled in the randomized cohort at any single investigational site.

Randomized Cohort:

Up to 300 subjects who meet all eligibility criteria will be randomized 2:1 by permuted block method (stratified by site and adjunctive lesion preparation) to one of two treatment arms:

* Intervention - treatment with SELUTION SLR™ 018 DEB
* Control - treatment with commercially available PTA (uncoated balloon)

Pharmacokinetic (pK) Sub-study:

The pK substudy is a parallel registry consisting of up to 20 additional consecutive subjects meeting all eligibility criteria treated with the SELUTION DEB recruited at select study sites. The separate PK substudy protocol details the schedule of evaluations and blood draws to characterize the pK plasma profile of sirolimus.

ELIGIBILITY:
Clinical Inclusion Criteria:

1. Subject age is ≥ 18 years or minimum legal age as required by local regulations.
2. Life expectancy >1 year in opinion of investigator.
3. Documented ischemia with Rutherford classification category 2, 3 or 4.
4. Target lesion(s) in the SFA or PPA.
5. Able to walk without the assistance of a walker.
6. Subject is willing and able to provide informed consent and comply with study procedures and required follow-up evaluations.
7. Female subjects only: If female, then subjects of childbearing potential must have a negative pregnancy test ≤ 7 days before the procedure and be prepared to use effective contraception for 12 months after treatment.

Angiographic Inclusion Criteria:

1. Angiographic evidence that target lesion lies within the superficial femoral artery and/or proximal popliteal artery (P1 and P2 only).
2. Angiographic evidence that the target lesion consists of either a de novo lesion or a non-stented restenotic lesion, or a combination of both, that meets one of the following criteria:

   A. A stenosis of 70-99% with lesion length between ≥3cm and <20cm by visual estimation.

   B. A total (100%) occlusion with lesion length between ≥3cm and ≤10cm by visual estimation.

   C. A combination lesion (stenosis and total occlusion) must have a total lesion length between ≥3cm and <20cm by visual estimation with an occluded segment that is ≤10cm by visual estimation.

   D. If multiple lesions are to be treated, then only 2 lesions may be included. The total combination of lengths must be between ≥3cm and < 20cm by visual estimation, and there must be at least 5 cm of artery that is not to be treated between them.
3. Target vessel reference diameter ≥4mm and ≤7mm.
4. Patent arterial inflow (common iliac, external iliac, common femoral and profunda femoris arteries, and the proximal 2 cm of the SFA) free from significant lesion (defined as ≥50% stenosis) as confirmed on angiography.

   Note: Where required, inflow iliac arteries (common and external iliac arteries only) must be successfully treated during the index procedure. Completion angiography must confirm successful treatment of inflow disease (≤30% residual stenosis, no distal embolization, and no Grade C or greater dissection ) prior to pre-dilation and randomization of the target lesion(s). Drug-eluting devices are not allowed for treatment of the occluded inflow iliac arteries.
5. Angiographic evidence of adequate distal run off (defined as ≤50% stenosis) in one or more tibial arteries on initial angiography, and if applicable, after completion of inflow artery treatment.

Note: Treatment of outflow disease is permitted during the index procedure. Drug-eluting devices are not allowed for outflow treatment.

PK Sub-Study Inclusion Criteria:

Subjects must meet all of the main protocol inclusion criteria to participate in the PK sub-study. Subjects must also meet the following additional PK sub-study inclusion criteria:

1. Subject is willing and able to provide informed consent for the PK sub-study and comply with the PK sub-study procedures and required follow-up evaluations.

Clinical Exclusion Criteria:

1. Other surgical or endovascular procedure in the target limb that occurred within 14 days prior to index procedure or is planned for within 30 days following index procedure, with exception for diagnostic angiography.
2. Inability to tolerate dual antiplatelet therapy.
3. Known hypersensitivity or allergy to Sirolimus or other pharmacologic agents, such as contrast agent, which are required for the procedure and which cannot be adequately pre-treated.
4. Stroke or MI within 3 months of enrollment.
5. Symptom onset less than 14 days prior to index procedure (acute limb ischemia).
6. Lower limb disease in the contralateral leg that requires treatment at the index procedure, or, that is planned within 14 days prior to the index procedure or within 30 days after the index procedure.
7. Prior vascular surgery (including bypass and endarterectomy) of abdominal aorta, iliac arteries, or arteries of the index limb.
8. Non-atherosclerotic disease of the index limb (including aneurysmal disease, vasculitis, Buerger's disease)
9. Target lesion requires treatment with alternative therapies such as thrombolysis, thrombus aspiration, cutting/scoring/contoured balloon, stenting, laser, cryoplasty, intravascular lithotripsy, brachytherapy, re-entry device).
10. Subject has target lesion(s) that require treatment via pedal site.
11. Subject has target lesion(s) that require access via upper extremity arteries.
12. Hypercoagulable state or disorder present, or coagulopathy present, including platelet count less than 80,000 per microliter.
13. Chronic renal insufficiency (dialysis dependent, or serum creatinine >2.5 mg/dL within 30 days of index procedure).
14. Systemic infection (WBC > 12,000 and febrile) or known immune compromise.
15. Breast-feeding woman.
16. Currently participating in another investigational drug or device study that has not completed primary endpoint follow-up.

Angiographic Exclusion Criteria:

1. Presence of a previously placed stent in the treated artery.
2. Failure to successfully cross the target lesion.
3. Residual stenosis ≥30% after pre-dilatation.

PK Sub-Study Exclusion Criteria:

1. Subjects must meet none of the main protocol exclusion criteria (Section 6.1.2 of the main protocol) to participate in the PK sub-study. Subjects will be excluded if any of the following additional PK sub-study exclusion criteria are met:
2. Any limus family (Zotarolimus, Everolimus, Sirolimus etc.) eluting device has been placed/used in any part of the body within 3 months prior to the index procedure including non-target lesion(s) treated during the index procedure.
3. Planned intervention with any limus family (Zotarolimus, Everolimus, Sirolimus etc.) eluting device anywhere in the body within 6 months after the index procedure. Note: staged procedures >30 days after index procedure (Exclusion #20 and #22 of the main protocol) are permitted only in the main protocol, and are not permitted in this PK sub-study.
4. The subject is taking or has taken within the last 3 months any limus family medication(s) for any reason.
5. Subjects who are taking strong CYP3A4 Inhibitors within 14 days before the index procedure or plan to take the strong inhibitors during the study period. Strong inhibitors include: cobicistat; ritonavir; indinavir and ritonavir; itraconazole; ketoconazole; lopinavir and ritonavir; paritaprevir and ritonavir and ombitasvir (and/or dasabuvir); posaconazole; saquinavir and ritonavir; tipranavir and ritonavir; elvitegravir and ritonavir; telithromycin; voriconazole; ceritinib; clarithromycin; idealalisib; nefazodone; nelfinavir.
6. Subjects who are taking strong CYP3A4 Inducers within 14 days before the index procedure or plan to take the strong inducers during the study period. Strong inducers include apalutamide; carbamazepine; enzalutamide; ivosidenib; lumacaftor and ivacaftor; mitotane; phenytoin; rifampin; St. John's wort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-06-24 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint | 12 months
  Primary patency of the target lesion defined as freedom from ANY of the following adverse events:
  * Clinically driven target lesion revascularization (CD-TLR, defined as re-intervention of target lesion(s) due to recurrent, persistent, or worsening symptoms and angiographic restenosis (≥ 50% diameter stenosis) of target lesion by ACL measurement) OR
  * Restenosis as determined by core lab adjudicated duplex ultrasound peak systolic velocity ratio of >2.4 or occlusion of the target lesion.
Primary Safety Endpoint | 30 days or 12 months
  The primary safety endpoint is the freedom from ANY of the following adverse events:
  * All-cause perioperative death (POD) [evaluated at 30 days] OR
  * Target limb major (above-the-ankle) amputation [evaluated at 12 months] OR
  * Clinically driven target lesion revascularization (CD-TLR) [evaluated at 12 months]
PK Sub-Study Primary Endpoint: C(max) | 6 months
  PK parameters of C(max).
PK Sub-Study Primary Endpoint: T(max) | 6 months
  PK parameters of T(max).
PK Sub-Study Primary Endpoint: AUC(last) | 6 months
  PK parameters of AUC(last).
PK Sub-Study Primary Endpoint MRT(last) | 6 months
  PK parameters of Mean Residence Time(last).

SECONDARY OUTCOMES:
Powered Secondary Endpoints | 12 months
  If both primary endpoints are met, the following endpoint will be tested for superiority in a sequential manner:
  • Clinically driven target lesion revascularization (CD-TLR)
Device success | Immediately following the procedure
  A secondary performance endpoint defined as successful delivery, balloon inflation, deflation, and retrieval of the intact investigational device.
Procedural (technical) success | Immediately following the procedure
  A secondary performance endpoint defined as device success and residual diameter stenosis ≤ 30% on completion angiography by core lab assessment.
Clinical success | Discharge defined as immediately prior to hospital discharge from the index procedure or within 7 days, whichever occurs first
  A secondary performance endpoint defined as procedural success without procedural complications (death, above-ankle target limb amputation, thrombosis of the target lesion or TLR) prior to discharge.
Secondary Safety Endpoints | 1, 6, and 12 months, and 2-5 years
  * Major adverse limb events (MALE).
  * Major cardiovascular events, myocardial infarction (MI), and stroke.
  * All-cause mortality.
Primary sustained clinical improvement | 1, 6, and 12 months, and 2-5 years
  A secondary efficacy endpoint defined as freedom from target limb major amputation and CD-TLR AND increase in Rutherford category from baseline.
Secondary sustained clinical improvement | 1, 6, and 12 months, and 2-5 years
  A secondary efficacy endpoint defined as freedom from target limb major amputation AND increase in Rutherford category from baseline.
  * Major amputation, defined as above-the-ankle amputation of the target limb.
  * Amputation-free survival, defined as freedom from all-cause mortality and major amputation.
Major amputation | 1, 6, and 12 months, and 2-5 years
  A secondary efficacy endpoint defined as above-the-ankle amputation of the target limb.
Amputation-free survival | 1, 6, and 12 months, and 2-5 years
  A secondary efficacy endpoint defined as freedom from all-cause mortality and major amputation.
Primary assisted patency | 12 and 24 months
  A secondary efficacy endpoint defined as freedom from target lesion occlusion by duplex ultrasound core laboratory [DCL] adjudication), irrespective of interventions for stenoses.
Secondary patency | 12 and 24 months
  A secondary efficacy endpoint defined as freedom from permanent occlusion (occlusion at the last follow-up imaging) as determined by the DCL.
  * Freedom from CD-TLR and binary restenosis as determined by the DCL [at 1, 3, 6, 12, 24, 36 months].
  * Any TLR, defined as any re-intervention of target lesion(s) 1, 6, and 12 months, and 2-5 years
Freedom from CD-TLR and binary restenosis | 1, 3, 6, 12, 24, 36 months
  A secondary efficacy endpoint defined as freedom from Clinically driven target lesion revascularization and binary restenosis as determined by the duplex ultrasound core laboratory (DCL).
Any TLR | 1, 6, and 12 months, and 2-5 years
  A secondary efficacy endpoint defined as any re-intervention of target lesion(s).
CD-TLR | 1, 6, and 12 months, and 2-5 years
  A secondary efficacy endpoint defined as re-intervention of target lesion(s) due to recurrent/persistent/worsening symptoms and the angiographic finding of ≥ 50% restenosis of target lesion by ACL measurement.
Clinically driven Target Vessel Revascularization (TVR) | 1, 6, and 12 months, and 2-5 years
  A secondary efficacy endpoint defined as re-intervention of target vessel due to recurrent/persistent/worsening symptoms and the angiographic finding of ≥ 50% restenosis of target vessel by ACL measurement.
Target lesion thrombosis | 1, 6, and 12 months, and 2-5 years
  A secondary efficacy endpoint assessed by angiographic or DUS core laboratory adjudication.
Rutherford category | 1, 6, 12, 24 and 36 months
  A secondary efficacy endpoint defined as change in Rutherford category from baseline.
Ankle brachial index (ABI) | 12 and 24 months
  A secondary efficacy endpoint defined as change in ankle brachial index (ABI) from baseline.
Walking capacity | 1, 6, 12, 24 and 36 months
  A secondary efficacy endpoint defined as change in Walking capacity assessed by Walking Impairment Questionnaire (WIQ) from baseline.
Secondary Imaging endpoints (DCL adjudicated): | 12 and 24 months
  * Primary duplex-defined binary restenosis - Peak Systolic Velocity Ratio (PSVR)>2.4.
  * Alternate duplex-defined binary restenosis - Peak Systolic Velocity Ratio (PSVR)>3.4.
Secondary Quality of life and health economic assessments (1) | 12 months
  • Change in EQ-5D score from baseline. OBS.: Following EuroQol terminology: Scores are anchored at 1 (full health) and 0 (a state as bad as being dead) as required by their use in economic evaluation. Values less than 0 represent health states regarded as worse than a state that is as bad as being dead.
Secondary Quality of life and health economic assessments (2) | 12 months
  • Days of target lesion-related hospitalization at 12 months.
PK Sub-Study Secondary Endpoint: AUC(inf) | 6 months
  If calculations are valid, additional PK parameter of AUC(inf).
PK Sub-Study Secondary Endpoint: Cl | 6 months
  If calculations are valid, additional PK parameter of Cl.
PK Sub-Study Secondary Endpoint: Vz | 6 months
  If calculations are valid, additional PK parameter of Vz.
PK Sub-Study Secondary Endpoint: Vss | 6 months
  If calculations are valid, additional PK parameter of Vss.
PK Sub-Study Secondary Endpoint: half-life | 6 months
  If calculations are valid, additional PK parameter of half-life.
PK Sub-Study Secondary Endpoint: C(max) | 6 months
  Dose normalized C(max) will be considered if appropriate.
PK Sub-Study Secondary Endpoint: AUC | 6 months
  Dose normalized AUC will be considered if appropriate.

CONTACTS AND LOCATIONS:
Locations (38):
- United States (28):
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Mission Cardiovascular Research Institute, Fremont, California
  - St. Helena Hospital, St. Helena, California
  - ClinRé, Thornton, Colorado
  - Vascular Care Group, Darien, Connecticut
  - Manatee Memorial Hospital, Bradenton, Florida
  - The Cardiac and Vascular Institute Research Foundation, Gainesville, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Palm Vascular Centers, Miami Beach, Florida
  - Guardian Research Organization, LLC, Winter Park, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Cardiovascular Consultants of South Georgia, Thomasville, Georgia
  - Heart Care Centers Research Foundation, Palos Park, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Cardiovascular Institute of the South, Gray, Louisiana
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Mercy Hospital, St Louis, Missouri
  - Holy Name Medical Center, Teaneck, New Jersey
  - James J. Peters VA Medical Center, The Bronx, New York
  - NC Heart and Vascular Research, LLC, Raleigh, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Miriam Hospital, Providence, Rhode Island
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
  - El Paso Cardiology, El Paso, Texas
  - Baylor College of Medicine, Houston, Texas
  - Heart Hospital Baylor Plano, Plano, Texas
  - Texas Cardiac and Vascular Institute San Antonio, San Antonio, Texas
- Universitätsklinikum Graz, Graz, Austria
- Germany (7):
  - Alexianer Klinikum Hochsauerland, Arnsberg
  - Universitäts-Herzzentrum Freiburg - Bad Krozingen, Bad Krozingen
  - Krankenhaus Buchholz, Buchholz
  - Sana Kliniken Oberfranken Coburg, Coburg
  - Universitätsklinikum Leipzig, Leipzig
  - RoMed Klinikum Rosenheim, Rosenheim
  - University Clinic Tübingen, Tübingen
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong, Pok Fu Lam
  - The Chinese University of Hong Kong, Shatin

IPD SHARING:
Plan to Share IPD: No